CLINICAL TRIAL: NCT00229359
Title: Risk Factors for PTSD
Brief Title: Characteristics of Post-Traumatic Stress Disorder (PTSD) and Non-PTSD Subjects
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-99-1813-JZ-CTIL
Record Dates: First submitted 2005-09-28; First posted 2005-09-29 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

SUMMARY:
Compare PTSD and non-PTSD subjects on several demographic, cognitive and military variables

ELIGIBILITY:
Inclusion Criteria:

* Subjects applied for treatment in the MOH rehabilitation centers or the IDF unit for combat reactions and were diagnosed with PTSD

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult
Dates: Start 2000-01; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zohar, MD, Principal Investigator — Tel Aviv University

REFERENCES:
- [Derived] Zohar J, Fostick L, Cohen A, Bleich A, Dolfin D, Weissman Z, Doron M, Kaplan Z, Klein E, Shalev AY; Israeli Consortium on PTSD. Risk factors for the development of posttraumatic stress disorder following combat trauma: a semiprospective study. J Clin Psychiatry. 2009 Dec;70(12):1629-35. doi: 10.4088/JCP.08m04378blu. Epub 2009 Oct 20. PMID 19852906